CLINICAL TRIAL: NCT01441765
Title: Phase II Study of PD-1 Blockade Alone or In Conjunction With the Dendritic Cell (DC)/Renal Cell Carcinoma (RCC) Fusion Cell Vaccination
Brief Title: PD-1 Alone or With Dendritic Cell/Renal Cell Carcinoma Fusion Cell Vaccine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Avigan, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-178; P50CA101942-06A1 (NIH)
Record Dates: First submitted 2011-09-22; First posted 2011-09-28 (Estimated); Results first posted 2016-11-09 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Renal Cell Carcinoma
Keywords: Kidney; Metastatic; Stage IV
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-011 (Active Comparator): CT-011 3 mg/kg for 4 cycles of 6 weeks
  Interventions: Drug: CT-011
- CT-011 with DC/RCC fusion vaccine (Active Comparator): CT-011 with DC/RCC fusion vaccine for subjects undergoing nephrectomy, resection of tumor tissue, or aspiration of malignant effusion
  Interventions: Drug: CT-011; Biological: DC/RCC fusion vaccine

INTERVENTIONS:
Drug: CT-011 — CT-011 at 3 mg/kg IV for 4 cycles of 6 weeks
Biological: DC/RCC fusion vaccine — Vaccination once per cycle on Day 8 of treatment cycles 2-4
  Arms: CT-011 with DC/RCC fusion vaccine

SUMMARY:
CT-011 is an investigational monoclonal antibody. Monoclonal antibodies are a type of drug that are known to target specific cells (in this case, cells in the immune system) The DC RCC Vaccine is agent that tries to help the immune system to recognize and fight against cancer cells.

The purpose of this research study is to determine the safety of CT-011 alone, and in combination with the Dendritic Cell Renal Cell Carcinoma (DC RCC) vaccine. The investigators are also trying to find out what effect the combination has on the disease, and on your immune system.

DETAILED DESCRIPTION:
This study is divided into 2 groups. The first 22 subjects will be in Group 1 and will receive CT-011 only. The next 22 subjects will be in Group 2 and will receive CT-011 and the DC RCC vaccine.

Group 1: Subjects in this cohort are not required to have tumor resection (nephrectomy) to participate in this study. For subjects who are undergoing nephrectomy and for subjects undergoing resection for another metastasis, infusions of CT-011 will begin 21 to 35 days post-surgery. Subjects will receive 4 cycles of CT-011 therapy. Each cycle consists of a dose of CT-011 given on days 1, 14, and 28 intravenously.

For subjects who are not undergoing nephrectomy for standard of care therapy, infusions of CT-011 will begin 21 to 28 days following registration on the study. Subjects will receive a total of four cycles of CT-011 therapy. Each cycle consists of a dose of CT-011 given on days 1, 14, and 28 intravenously.

Group 2: Subjects in this cohort will have chosen to undergo a "debulking nephrectomy" (surgery to remove a tumor of the kidney, but not all of the cancer cells in your body) as a standard treatment for kidney cancer or have tumor lesions that are accessible (may be removed without major surgery) and are being removed to treat or diagnose their cancer. All subjects in this group will receive infusions of CT-011 21 to 35 days following tumor resection.

Subjects will receive a total of 4 cycles of CT-011 therapy. Each cycle consists of a dose of CT-011 given on days 1, 14, and 28. In addition they will receive a vaccination of the DC RCC vaccine on day 8 of each cycle.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV renal cancer
* Measurable disease
* Life expectancy > 3 months
* Adequate organ and marrow function

Exclusion Criteria:

* Clinical evidence of central nervous system (CNS) disease. Subjects with a history of treated brain metastasis must be stable with no evidence of disease for 3 months
* Clinically significant autoimmune disease
* HIV+
* Serious intercurrent illness such as infection requiring intravenous (IV) antibiotics, or significant cardiac disease characterized by significant arrhythmia, uncontrolled hypertension, unstable ischemic coronary disease or congestive heart failure
* Pregnant or lactating
* History of clinically significant venous thromboembolism (For Cohort 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Started | 11 | 0 (not opened)
Completed | 10 | 0 (not opened)
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine | Total
Number analyzed (Participants) | 11 | 0 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 6 |  | 6
  >=65 years | 5 |  | 5
Age, Continuous [Mean (Full Range); unit: years] | 63 [43 to 78] |  | 63 [43 to 78]
Gender [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 8 |  | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 |  | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Assessment of toxicity associated with treating patients with metastatic RCC with CT-011 alone or CT-011 in conjunction with DC/RCC. Toxicity was assessed and classified according to CTCAE Version 4.0.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Number analyzed (Participants) | 10 | 0
participants | 8 |

2. Primary Outcome: Number of Participants With PR or CR at 2 Years
Description: To evaluate the complete and partial response rate following completing 4 cycles of CT-011 alone or CT-011 in conjunction with DC/RCC fusion vaccine. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, (with an absolute increase of at least 5 mm), or the appearance of new lesions. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study."
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Number analyzed (Participants) | 10 | 0
participants | 0 |

3. Secondary Outcome: Immunologic Response
Description: To evaluate immunologic response directed against RCC and tumor specific antigens following therapy with CT-011 alone or CT-011 in conjunction with DC/RCC fusion vaccine. Immunologic response will be characterized as peak response post-therapy and ongoing response at 3 and 6 months following treatment.
Time Frame: 2 years
Population: Data was not analyzed as so few participants were enrolled and none of the participants achieved a PR or CR.
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Effect on Circulating Regulatory T Cells
Description: To evaluate the effect of CT-011 alone or in conjunction with DC/RCC fusions on circulating regulatory T cells and PD-1 expression by circulating and bone marrow derived T cells.
Time Frame: 2 years
Population: Data was not analyzed as so few participants were enrolled and no participants achieved a PR.
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Who Survived at 2 Years
Description: To evaluate overall survival following treatment with CT-011 alone or CT-011 in conjunction with DC/RCC fusion vaccine.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Number analyzed (Participants) | 10 | 0
participants | 4 |

ADVERSE EVENTS:
Arm/Group | CT-011 | CT-011 With DC/RCC Fusion Vaccine
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 8/10 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-011 (N=10) | CT-011 With DC/RCC Fusion Vaccine (N=0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0
Flatulence (Gastrointestinal disorders) | 1 (1) | 0
Neutropenia (Investigations) | 1 (1) | 0
Hyperkalemia (Investigations) | 1 (1) | 0
Hypothyroidism (Investigations) | 2 (3) | 0
Weight Loss (Metabolism and nutrition disorders) | 1 (1) | 0
Pneumonitis (General disorders) | 1 (1) | 0
Pruritis (Investigations) | 1 (1) | 0
Fever (General disorders) | 1 (1) | 0
Rash (back/neck) (General disorders) | 1 (1) | 0
Cough (Investigations) | 1 (1) | 0

LIMITATIONS AND CAVEATS:
Due to lack of funding, the study was terminated early without completing enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No